CLINICAL TRIAL: NCT04188808
Title: A Prospective Case-control Study of the Quality of Life in Patients With Aneurysmatic or Occlusive Disease in the Lower Limb
Brief Title: Prospective Case-control Study in Patients With PAA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rebecka Hultgren (Other)
Collaborators: Karolinska University Hospital (Other); Karolinska Institutet (Other); Stockholm South General Hospital (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Rebecka Hultgren, Principal Investigator, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NPAA0831365
Record Dates: First submitted 2019-11-13; First posted 2019-12-06 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Popliteal Artery Aneurysm; Peripheral Arterial Disease; Quality of Life
Keywords: Open vascular surgery; Vascular disease
MeSH Terms: conditions — Popliteal Artery Aneurysm; Peripheral Arterial Disease; Vascular Diseases | interventions — Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Popliteal artery aneurysm (Experimental): Asymptomatic popliteal artery aneurysm patients will undergo surgery with a femoropopliteal/femorodistal bypass
  Interventions: Other: Bypass surgery
- Peripheral artery disease (Active Comparator): Patients with peripheral artery disease defined as (ankle - brachial index, ABI <0.5 or typical symptoms); intermittent claudication (IC), or resting pain and/or minor tissue loss. Will undergo surgery with a femoropopliteal/femorodistal bypass
  Interventions: Other: Bypass surgery

INTERVENTIONS:
Other: Bypass surgery — All patients scheduled for elective surgery of PAA and PAD.

SUMMARY:
The overall objective is to highlight different aspects of care in patients with PAA before and after treatment, and identifying factors that influence the outcome of PAA patients.

DETAILED DESCRIPTION:
An aneurysm is most commonly defined as a permanent focal dilatation of an artery to 1.5 times its normal diameter. While the abdominal aorta is the most common site of aneurysm formation, the popliteal artery (PA) represents the second most common site of aneurysm formation, accounting for more than 70 percent of all peripheral aneurysms. A popliteal artery aneurysm (PAA) is a focal dilatation of the popliteal artery (red arrow). PAAs are rare in the general population but more commonly found in patient populations with other aneurysms, such as abdominal aortic aneurysm (AAA). Within the general population, PAAs are predominantly found in men and are extremely rare in women. There are few studies on the prevalence of PAAs in healthy individuals, but 14-19% of male and 12% of female AAA patients have PAAs. There is no clear correlation between the diameter of the AAA and the prevalence of PAA. There is furthermore a lack of consensus of the precise arterial diameter that defines a PAA.

It is paramount to identify and treat PAA patients before acute symptoms develop, given the high risk of major complications associated with acute presentation, such as major amputation. Unfortunately, there is a lack of knowledge of the natural history for PAAs, which is why surgical procedures are recommended mainly based on clinical experience and guidelines developed from insufficient scientific information. The preventive purpose, more specifically to prevent the risk of acute symptom development, should be evaluated against the frequency of complications inflicted by surgical treatment, so called "surgical risk". For this reason, it is important to evaluate the patients' health-related quality of life (HRQoL) before and after treatment in order to determine how the surgical treatment affect patients. In general, the Health-Related Quality of Life (HRQoL) is therefore emerging as an important outcome measure for interventions designed to improve patient's health, well-being, or both. There is very limited prior knowledge of HRQoL outcomes following surgical treatment of PAAs and the PAA patient's HRQoL, and whether-and to what extent- it becomes affected by the surgical treatment, is yet unknown. The surgical treatment in PAA patients and patients with peripheral arterial disease (PAD), are comparable whereas the underlying pathologies are distinct. Thus, peripheral arterial disease patients commonly experience substantial symptom relief following a surgical intervention (i.e. lower limb pain is alleviated, or ischemic wound healing is promoted). By contrast, PAA patients are often asymptomatic prior to surgery. It is therefore conceivable that a surgical intervention in PAA patients translates to a lower HRQoL after surgery than what is observed following bypass surgery for PAD. However, this needs to be further explored and confirmed in prospective studies.

Aim To investigate whether the QoL of PAA patients compared to PAD patients after surgical and potential changes over time.

Hypothesis Compared to PAD patients, femoropopliteal/femorodistal bypass surgery interventions undertaken on PAA patients result in a more pronounced negative HRQoL impact.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for elective surgery of PAA (asymptomatic)
* All patients scheduled for elective surgery of PAD
* Elective open surgery
* Intermittent claudication
* Resting pain or very limited minor tissue loss

Exclusion Criteria:

* Cognitive failure
* Major tissue loss
* severe pain
* if one cannot assimilate information in Swedish and understand the questionnaires

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
SF-36 | Five years
  A 36-item questionnaire that measures 8 dimensions of physical and mental health. ( 0-100) Positive if high

SECONDARY OUTCOMES:
EQ-5D | Five years
  EQ-5D is a standardized instrument for measuring generic health status (0-100) 100 best Health and 0 worst helath

OTHER OUTCOMES:
PHQ-9 PHQ-9 | Five years
  Depressive symptoms were assessed with the validated nine-item. Patient Health Questionnaire. The PHQ provides a dichotomous measure of depressive symptoms ( 0- 30; below 4 = no deression; 10 or above = depression)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecka Hultgren, Prof, Principal Investigator — Karolinska Instutet
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No